CLINICAL TRIAL: NCT05597189
Title: Clinical Study of Palliative / Preventive Treatment of Chronic Back Pain by Taking a Dietary Supplement Based on Botanical Extracts
Brief Title: Clinical Study for Palliative/Preventive Treatment of Chronic Back Pain
Acronym: Backin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: UCAMCFE-00028
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2022-09

CONDITIONS: Supplementation; Back Pain
Keywords: botanical extracts
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botanical extracts high dose (Experimental): Consumption for 84 days. Subjects should consume two capsules half an hour before breakfast.
  Interventions: Dietary Supplement: Experimental product
- Botanical extracts low dose (Experimental): Consumption for 84 days. Subjects should consume two capsules half an hour before breakfast.
  Interventions: Dietary Supplement: Experimental product
- Control group (Placebo Comparator): Consumption for 84 days. Subjects should consume two capsules half an hour before breakfast.
  Interventions: Other: Control product consumption

INTERVENTIONS:
Dietary Supplement: Experimental product — Botanical extract
  Arms: Botanical extracts high dose; Botanical extracts low dose
Other: Control product consumption — Product with identical characteristics to the experimental product.
  Arms: Control group

SUMMARY:
Randomized, controlled, double-blind, double-blind clinical trial, with three parallel arms depending on the product consumed (experimental product dose 1 and dose 2 and placebo product) and single-center, to measure the efficacy of a botanical supplement on the prevention of non-joint pain.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will be randomly assigned to each of the study groups (investigational product dose 1 or dose 2, or placebo, depending on the group to which they have been assigned).

The product to be consumed is a Botanical Extract. Participants will consume the product for 84 days. It should be taken half an hour before breakfast, two capsules per day.

The study subjects will have to make 5 visits to the laboratory. On the first and last visit, they will have their blood drawn, their sleep quality will be evaluated and they will complete a series of questionnaires to evaluate their quality of life and type of back pain. In the rest of the visits they will only have to take the tests on paper.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 and 65 years of age.
* The subjects must have localized myofascial pain in the back area (cervical, dorsal and lumbar), with an evolution time of at least 3 months.
* The pain must present an initial score of at least 30 mm in the pain evaluation by means of the VAS scale.
* The pain must be episodic.
* BMI 18.5 - 29.9 kg/m2.
* Subjects should not be treated with narcotic drugs or steroidal anti-inflammatory drugs. steroidal anti-inflammatory drugs or immunosuppressants.

Exclusion Criteria:

* Severe or terminal illnesses.
* Subjects with pain associated with trauma.
* Subjects with pain associated with chronic conditions (rheumatoid arthritis, herniated discs, ankylosing herniated disc, ankylosing spondylitis, etc.).
* Subjects with known allergy to any of the components of the investigational product. the investigational product.
* Subjects undergoing physiotherapy treatment during the course of the study. development of the study.
* Pregnant or lactating women.
* Inability to understand the informed consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain from baseline at 12 weeks | The evolution of pain after consumption during 12 weeks will be measured.
  Visual analog scale from 0 to 10. The higher the value, the more pain.

SECONDARY OUTCOMES:
Change in concomitant analgesic medication | The test will be measured at baseline and after 12 weeks of consumption. It will also be evaluated on a daily basis
  The change in the need for the use of analgesic medications will be evaluated
Evaluation of back pain: Promis-29 test | Day 1, at 4, 8 and 12 weeks later
  Back pain will be measured with the Promis-29 v2.0 test. This is a 29-item test that measures the degree of pain.
Evaluation of back pain: Cornell | Day 1, at 4, 8 and 12 weeks later
  The Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) assesses musculoskeletal symptomatology in workers who perform sedentary and standing work. sedentary work and standing work.
Level of functionality: Roland Morris test | Day 1, at 4, 8 and 12 weeks later
  The Roland-Morris questionnaire is used to reliably determine the degree of physical degree of physical disability derived from non-specific low back pain.
Quality of life questionnaire | Day 1, at 4, 8 and 12 weeks later
  SF-36 test health questionnaire
Wellbeing / wellness | Day 1, at 4, 8 and 12 weeks later
  WHOQOL BREF test
Depression | Day 1, at 4, 8 and 12 weeks later
  Beck depression. Test to measure the level of depression of the subjects
Anxiety questionnaire | Day 1, at 4, 8 and 12 weeks later
  Test STAI, to measure the level of anxiety of the subjects
Perceived stress | Day 1, at 4, 8 and 12 weeks later
  Remor, 2001. Test to measure the level of stress of the subjects
Sleep quality | It will be measured twice, once at baseline or at the end of the study after 12 weeks of use
  Measured by Pittsburgh test
Body composition | The test will be measured at baseline and after 12 weeks of consumption.
  It is a control variable. Measured by bioimpedance
Physical activity | The test will be measured at baseline and after 12 weeks of consumption. It will be measured during 3 weekdays and one weekend day.
  It is a control variable. Measured by accelerometry, with Actigraph wGT3X-BT
Sleep efficiency | The test will be measured at baseline and after 12 weeks of consumption. It will be measured during 3 weekdays and one weekend day.
  Measured by accelerometry, with Actigraph wGT3X-BT
C Reactive Protein (PCR) | It will be measured twice, once at baseline or at the end of the study after 12 weeks.
  It is a blood test that measures inflammation levels.
Interleukin 6 (IL-6) | It will be measured twice, once at baseline or at the end of the study after 12 weeks.
  It is a blood test that measures inflammation levels.
Liver safety variables | It will be measured twice, once at baseline or at the end of the study after 12 weeks.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain